CLINICAL TRIAL: NCT02350179
Title: Efficacy of Tranexamic Acid in Reducing Blood Loss During and After Caesarean Section
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Zarafshan Mohammad Raqeeb, Student, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ASU1115
Record Dates: First submitted 2015-01-01; First posted 2015-01-29 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Hemorrhage of Cesarean Section and/or Perineal Wound
MeSH Terms: interventions — Tranexamic Acid; Glucose

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cases (Experimental): Women assigned to the study group will receive 1 gr of Tranexamic acid injection (Kapron, AMOUN Pharmaceutical co.) given slowly I.V over 10 minutes before the operation.
  Interventions: Drug: Tranexamic Acid
- control (Placebo Comparator): The control group will receive 30ml of 5% glucose. Both provider and patient will be double-blinded until the conclusion of the study.
  Interventions: Drug: Glucose

INTERVENTIONS:
Drug: Tranexamic Acid — This will be a prospective, randomized controlled trial that will be carried at Obstetrics and Gynecology Department, Ain Shams Maternity Hospital.
  The study will include 100 pregnant women with singleton fetus 38 or more weeks gestation who will be divided in to two groups.
  Study group will include 50 women and control group will include 50 women. Women assigned to the study group will receive 1 gr of TXA injection (Kapron, AMOUN Pharmaceutical co.) given slowly I.V over 10 minutes before the operation.
  The control group will receive 30ml of 5% glucose. Both provider and patient will be double-blinded until the conclusion of the study.
  Other Names: Efficacy of Tranexamic Acid
  Arms: cases
Drug: Glucose — The control group will receive 30ml of 5% glucose. Both provider and patient will be double-blinded until the conclusion of the study.
  Arms: control

SUMMARY:
The aim of this study is to evaluate the efficacy of tranexamic acid in reducing blood loss during and after elective C.S.

The Research Question Is Tranexamic acid effective in reducing blood loss during and after elective Caesarean section?

The Research Hypothesis The TXA could be able to reduce blood loss during and after elective Caesarean section.

The null hypothesis will therefore state that:

There will be no difference between TXA and placebo in reducing blood loss during and after elective Caesarean section.

DETAILED DESCRIPTION:
Caesarean Section (C.S) is the most common major surgical procedure performed on women worldwide and its rates continue to rise steadily in both developed and developing countries (Gibbons et al., 2012).

Caesarean Section is associated with more blood loss than vaginal delivery; there is a trend for increasing rates in both developed and developing countries (Betra´n, 2007).

The National US Caesarean section rate leveled off at 32.8% in 2010 and 2011 (Hamilton et al., 2012).

Caesarean Section accounts for 20-25% of all deliveries in the UK (Fairley Dundas, 2011).

C.S rates have increased to as high as 25-30 % in many areas of the world, in Pakistan the (C.S) rate is 25% (Najmi, 2000).

In many areas of China the (C.S) rate is as high as 40-50% (Zhang, 2008). The main causes of death following a (C.S) are infection, hemorrhage, pulmonary embolism, and anesthesia - associated complications, caesarean section has been an important underlying cause of death in Norway and contributed to the increased maternal death ratio in the last decade (Vangen and Bergsjo, 2003).

Delivery by (C.S) can cause more complications than normal vaginal delivery and one of the most common complications is primary or secondary postpartum hemorrhage up to 20% (Lu et al., 2005).

Obstetric hemorrhage can be life threatening, therefore to reduce the morbidity and mortality due to obstetric hemorrhage we need to reduce the bleeding at C.S (Bingham, 2012).

Postpartum hemorrhage is a major cause of maternal mortality, especially in under-resourced countries, accounting for nearly one - quarter of all maternal deaths worldwide (WHO, 2007). Recent studies from developed countries reported an increase in the rate of postpartum hemorrhage, which has been attributed (at least in part) to arise in the rate of C.S (Bateman et al., 2010).

As the incidence of Caesarean Section is increasing, and the average blood loss during Caesarean Section is (1000 ml) is double the amount of lost during vaginal delivery (500 ml) (Magann, 2005).

The hematocrit falls by 10 % and blood transfusion is required in 6% of woman undergoing Caesarean Section, Compared with 4% of woman who have a vaginal birth (RCOG, 2004).

Tranexamic acid (TXA) is a synthetic derivative of the amino acid lysine that exerts its anti-fibrin lytic effect through the reversible blockade of lysine binding sites on plasminogen molecules. It has been in used for many years for reducing the blood loss in surgeries (Astedt, 1987).

TXA has been shown to be very useful in reducing blood loss and incidence of blood transfusion in many surgeries.In gynecology and obstetrics, TXA is most commonly used to treat idiopathic menorrhagia and is an effective and well - tolerated treatment when administered orally. Bleeding associated with pregnancy (placental abruption, placenta previa) has also been treated with TXA (Dunn, 1999).

Furthermore, some randomized controlled studies have shown that TXA reduces blood loss after C.S (As et al., 1996).

No large randomized controlled trail of the efficacy of TXA in controlling blood loss during C.S has been reported, This randomized double blind, placebo controlled study will evaluates the efficacy of TXA in reducing blood loss during and after C.S.

Aim of the Work The aim of this study is to evaluate the efficacy of tranexamic acid in reducing blood loss during and after elective C.S.

The Research Question Is Tranexamic acid effective in reducing blood loss during and after elective Caesarean section?

The Research Hypothesis The TXA could be able to reduce blood loss during and after elective Caesarean section.

The null hypothesis will therefore state that:

There will be no difference between TXA and placebo in reducing blood loss during and after elective Caesarean section.

Patients and Methods This will be a prospective, randomized controlled trial that will be carried at Obstetrics and Gynecology Department, Ain Shams Maternity Hospital.

The study will include 100 pregnant women with singleton fetus 38 or more weeks gestation who will be divided in to two groups.

Study group will include 50 women and control group will include 50 women. Women assigned to the study group will receive 1 gr of TXA injection (Kapron, AMOUN Pharmaceutical co.) given slowly I.V over 10 minutes before the operation.

The control group will receive 30ml of 5% glucose. Both provider and patient will be double-blinded until the conclusion of the study.

The type of anesthesia will be decided by the surgeon and anesthetist after counseling the patient.

The inclusion criteria for the trial include:

* Pregnant women aged 20-40 with singleton fetus 38 or more weeks.
* Uncomplicated pregnancy, up to 3rd parity.
* Women undergoing scheduled elective C.S.

Exclusion criteria will include:

* Causes of uterine over-distention such as polyhydramnios or macrosomia
* Grand multi parity
* Previous PPH (3 x risk) or previous history of retained placenta
* Pre-eclampsia or pregnancy-induced hypertension
* Maternal hypertension.
* Pre-existing maternal hemorrhagic conditions
* Maternal diabetes mellitus.
* Abnormal placenta
* Sensitivity to TXA.
* Women taking anticoagulant therapy.

Assessment of the intraoperative blood loss will be started after the uterine incision by collection of the suctioned blood and by weighing surgical towels.

Post-operative blood loss will be assessed during the first 24 hour by weighingthe pads. HB level & Hematocrit will be investigated before and 24 hours after surgery.

The weight of the dry towels will be subtract from the weight of wet towels and the weight of the blood will be change in to volume using the formula {density of blood is 1060/m3; slightly denser then water so volume of the blood = weight multiply 0,9}).

Sample size determination:

Assuming a rate of intraoperative blood loss ranging between 650ml in group 1 & 450ml in group 2 with a SD of 300ml, a sample size of 48 patients in each group is enough to detect such difference, if true, at 0,05 alpha error and 0,09 power of the test (Kemal, 2010).

Randomization and allocation:

Interventional randomized controlled trial will be conducted using systemic random sampling allocation.

Dark sealed envelopes containing the intervention and taken from a table of numbers, created by a third party not involved in the allocation process.

Randomization will be performed by picking one envelope for each patient from sequentially numbered envelopes on the day of intervention initiation, by a nurse not involved in the study and the patient will informed about the allocation arm.

Blinding: This will be a randomized double blind trial, both the provider and researcher will be blinded to reduce bias; double-blind, placebo-controlled clinical trial, neither the provider nor the researchers know who is getting a placebo and who is getting the treatment to avoid information and calculation bias.

Ethical consideration and informed consent This clinical trial will be proposed to the ethical and review committee of Ain Shams University for approval.

An informed consent explaining the clinical trial and possible side effects of TXA will be obtained from each patient included in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 20-40 with singleton fetus 38 or more weeks
* Uncomplicated pregnancy, up to 3rd parity
* Women undergoing scheduled elective C.S

Exclusion Criteria:

* Causes of uterine over-distention such as polyhydramnios or macrosomia
* Grand multi parity
* Previous PPH (3 x risk) or previous history of retained placenta
* Pre-eclampsia or pregnancy-induced hypertension
* Maternal hypertension
* Pre-existing maternal hemorrhagic conditions
* Maternal diabetes mellitus
* Abnormal placenta
* Sensitivity to TXA
* Women taking anticoagulant therapy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Amount of blood loss calculated using statistical measurements to determine the total decrease in HB and Hematocrit levels following the CS | 6 months
  Assessment of the intra-operative blood loss will be started after the uterine incision by collection of the suctioned blood and by weighing surgical towels.
  Post-operative blood loss will be assessed during the first 24 hour by weighing the pads. HB level & Hematocrit will be investigated before and 24 hours after surgery.
  The weight of the dry towels will be subtracted from the weight of wet towels and the weight of the blood will change in to volume using the formula {density of blood is 1060/m3; slightly denser then water so volume of the blood = weight multiply 0,9}).
  Sample size determination:
  Assuming a rate of intraoperative blood loss ranging between 650ml in group 1 & 450ml in group 2 with a SD of 300ml, a sample size of 48 patients in each group is enough to detect such difference, if true, at 0,05 alpha error and 0,09 power of the test (Kemal, 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Zarafshan M Raqeeb, MS, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin: Clinical Management Guidelines for Obstetrician-Gynecologists Number 76, October 2006: postpartum hemorrhage. Obstet Gynecol. 2006 Oct;108(4):1039-47. doi: 10.1097/00006250-200610000-00046. PMID 17012482
- [Background] As AK, Hagen P, Webb JB. Tranexamic acid in the management of postpartum haemorrhage. Br J Obstet Gynaecol. 1996 Dec;103(12):1250-1. doi: 10.1111/j.1471-0528.1996.tb09638.x. No abstract available. PMID 8968245
- [Background] Astedt B. Clinical pharmacology of tranexamic acid. Scand J Gastroenterol Suppl. 1987;137:22-5. PMID 3321402
- [Background] Bateman BT, Berman MF, Riley LE, Leffert LR. The epidemiology of postpartum hemorrhage in a large, nationwide sample of deliveries. Anesth Analg. 2010 May 1;110(5):1368-73. doi: 10.1213/ANE.0b013e3181d74898. Epub 2010 Mar 17. PMID 20237047
- [Background] Betran AP, Merialdi M, Lauer JA, Bing-Shun W, Thomas J, Van Look P, Wagner M. Rates of caesarean section: analysis of global, regional and national estimates. Paediatr Perinat Epidemiol. 2007 Mar;21(2):98-113. doi: 10.1111/j.1365-3016.2007.00786.x. PMID 17302638
- [Background] Bingham D. Obstetric hemorrhage-related maternal mortality and morbidity. J Womens Health (Larchmt). 2012 Sep;21(9):901-2. doi: 10.1089/jwh.2012.3873. No abstract available. PMID 22928671
- [Background] Bick D; National Collaborating Centre for Women's and Children's Health; National Institute for Clinical Excellence. Caesarean Section. Clinical Guideline. National Collaborating Centre for Women's and Children's Health: commissioned by the National Institute for Clinical Excellence. Worldviews Evid Based Nurs. 2004;1(3):198-9. doi: 10.1111/j.1524-475X.2004.04060.x. No abstract available. PMID 17163898
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Lu MC, Fridman M, Korst LM, Gregory KD, Reyes C, Hobel CJ, Chavez GF. Variations in the incidence of postpartum hemorrhage across hospitals in California. Matern Child Health J. 2005 Sep;9(3):297-306. doi: 10.1007/s10995-005-0009-3. PMID 16132205
- [Background] Magann EF, Evans S, Hutchinson M, Collins R, Lanneau G, Morrison JC. Postpartum hemorrhage after cesarean delivery: an analysis of risk factors. South Med J. 2005 Jul;98(7):681-5. doi: 10.1097/01.SMJ.0000163309.53317.B8. PMID 16108235
- [Background] Najmi RS, Rehan N. Prevalence and determinants of caesarean section in a teaching hospital of Pakistan. J Obstet Gynaecol. 2000 Sep;20(5):479-83. doi: 10.1080/014436100434640. PMID 15512631
- [Background] Queenan JT. How to stop the relentless rise in cesarean deliveries. Obstet Gynecol. 2011 Aug;118(2 Pt 1):199-200. doi: 10.1097/AOG.0b013e3182266682. No abstract available. PMID 21775834
- [Background] Vangen S, Bergsjo P. [Do women die from pregnancy these days?]. Tidsskr Nor Laegeforen. 2003 Dec 23;123(24):3544-5. Norwegian. PMID 14691495
- [Background] Mathai M, Gulmezoglu AM, Hill S. Saving womens lives: evidence-based recommendations for the prevention of postpartum haemorrhage. Bull World Health Organ. 2007 Apr;85(4):322-3. doi: 10.2471/blt.07.041962. No abstract available. PMID 17546315
- [Background] Zhang J, Liu Y, Meikle S, Zheng J, Sun W, Li Z. Cesarean delivery on maternal request in southeast China. Obstet Gynecol. 2008 May;111(5):1077-82. doi: 10.1097/AOG.0b013e31816e349e. PMID 18448738